CLINICAL TRIAL: NCT06720311
Title: Comparison Between Modified Tubeless Super-Mini Percutaneous Nephrolithotomy, Flexible Ureterorenoscopy and Shockwave Lithotripsy for Treatment of Medium-sized Renal Stones: a Randomized Study
Brief Title: Management of Medium Sized Renal Stones
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Hamdan Gameel, Urologist, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AssiutU AGameel
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Renal Stones
Keywords: Medium sized renal stones
MeSH Terms: conditions — Nephrolithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Modified Tubeless Super-Mini Percutaneous Nephrolithotomy (Active Comparator)
  Interventions: Procedure: Modified Tubeless Super-Mini Percutaneous Nephrolithotomy
- Flexible Ureterorenoscopy (Active Comparator)
  Interventions: Procedure: Flexible Ureterorenoscopy
- Shockwave Lithotripsy (Active Comparator)
  Interventions: Procedure: Shockwave Lithotripsy

INTERVENTIONS:
Procedure: Modified Tubeless Super-Mini Percutaneous Nephrolithotomy — Modified Tubeless Super-Mini Percutaneous Nephrolithotomy
  Arms: Modified Tubeless Super-Mini Percutaneous Nephrolithotomy
Procedure: Flexible Ureterorenoscopy — Flexible Ureterorenoscopy
  Arms: Flexible Ureterorenoscopy
Procedure: Shockwave Lithotripsy — Shockwave Lithotripsy
  Arms: Shockwave Lithotripsy

SUMMARY:
Urinary stone disease is a common urological condition that affects millions of people worldwide, often leading to significant morbidity and healthcare costs. Medium-sized renal stones, typically defined as stones measuring 1 to 2 cm in diameter, pose a particular challenge in management. These stones are large enough to potentially cause significant obstruction and symptoms, yet their size and location make selecting an optimal treatment modality crucial for achieving favorable outcomes with minimal complications.

Historically, open surgery was the primary intervention for large or complex stones. However, the advent of minimally invasive techniques has revolutionized stone management, allowing for more effective and patient-friendly approaches. Among these, Super-mini percutaneous nephrolithotomy (SMP), flexible uretero-renoscopy (F-URS), and shock wave lithotripsy (SWL) have emerged as minimally invasive modalities for managing medium-sized renal stones.

This study aims to evaluate the outcomes; safety, efficacy, and complications associated with SMP versus F-URS Versus SWL in the management of reanl stones 10-20 mm in diameter.

DETAILED DESCRIPTION:
1. SWL All cases will be treated as day care procedures, under analgesia without any anesthesia. Dornier MedTech (Compact Delta II), an electromagnetic shock wave lithotripter will be used. Patients will be treated in supine position and the calculus will be localized by using X-ray or Ultrasound. All sessions will be performed by a single technician under the supervision of a urology consultant. Shock waves will be delivered at the rate of 60-80 per minute with a maximum of 2500 shocks per session of treatment. Session will be started with low energy waves and gradually increased according to patient tolerability. A maximum of 2 sessions spaced two weeks apart. All patients will be advised to drink lots of fluids and maintain active lifestyle and skipping exercises if possible. Prior to every sitting an X-ray KUB will be obtained to see for the state of clearance of stone.
2. Tubeless Super mini-PCNL (SMP) Modified technique will be performed in prone position using 14 Fr Amplatz sheath with the use of Karl Stroz semi rigid ureteroscope, Holmium Laser. Lithotripsy will be achieved by means of Holmium laser fiber 365 um.

   Ureteric catheter will be removed after 24 hours unless there is indications for JJ stent insertion ( eg. Only functioning kidney, perforation, etc)
3. F-URS A sensor guide wire was placed into the renal pelvis via rigid ureteroscope. A 11-13 Fr access sheath will be placed into the ureter, if possible. After ureteral access was obtained, a 8 Fr flexible ureteroscope will be used for the stone treatment. The stones disintegration by holmium laser fibers. At the end of the procedure, a ureteral stent (JJ stent or Ureteric catheter) will be inserted

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years old)
* Single renal stones 10-20 mm in longest dimension

Exclusion Criteria:

* Previous upper urinary tract exploration in ipsilateral side.
* Patients with JJ stent in ipsilateral side.
* Absolute contraindications to SWL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Stone free rate | 3 months
  1. SFR (by MSCT KUB) a patient is considered stone-free if the remaining fragments are less than 3 mm in size after 3 months of the procedure

IPD SHARING:
Plan to Share IPD: No